CLINICAL TRIAL: NCT04470622
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study of Aprepitant Injectable Emulsion in Early Hospitalized Adult Patients With COVID-19
Brief Title: Aprepitant Injectable Emulsion in Patients With COVID-19 (GUARDS-1)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated early by Heron, and was not terminated for safety reasons.
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HTX-019-202
Record Dates: First submitted 2020-07-13; First posted 2020-07-14 (Actual); Results first posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: COVID-19
Keywords: COVID-19; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group 1 (Experimental): Aprepitant injectable emulsion.
  Interventions: Drug: Aprepitant injectable emulsion
- Treatment Group 2 (Placebo Comparator): Saline placebo.
  Interventions: Drug: Saline Placebo

INTERVENTIONS:
Drug: Aprepitant injectable emulsion — Aprepitant injectable emulsion, once daily (QD) for 14 days.
  Arms: Treatment Group 1
Drug: Saline Placebo — Saline Placebo, once daily (QD) for 14 days.
  Arms: Treatment Group 2

SUMMARY:
The study will evaluate the efficacy and safety of aprepitant injectable emulsion added to standard of care for hospitalized patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Is hospitalized for ≤48 hours with SARS-CoV-2 infection. Confirmed by polymerase chain reaction (PCR), antigen or immunoglobulin M (IgM) antibody test.
* Has at least 1 of the following: Radiographic infiltrates by imaging, or oxygen saturation of <94% by pulse oximetry on room air or requiring supplemental oxygen.
* Not anticipated to require mechanical ventilation within 48 hours.

Exclusion Criteria:

* Is taking high-dose hydroxychloroquine or chloroquine.
* Is taking pimozide or strong or moderate CYP3A4 inhibitors.
* Is currently receiving treatment with products intended to modify immune response to COVID-19 (exception: dexamethasone, methylprednisolone, or equivalent are allowed), chemotherapy or on hemodialysis or peritoneal dialysis.
* Has known hypersensitivity to any components of aprepitant injectable emulsion.
* Has evidence of ARDS.
* Is being treated with oxygen delivered by high-flow nasal cannula nonrebreather mask, noninvasive positive pressure ventilation, or ECMO.
* Has multiple organ failure.
* Has current confirmed Influenza A or B infection, or a a history of organ or hematologic transplant, HIV, or active hepatitis B or hepatitis C infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-06-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Helen Keller Hospital, Sheffield, Alabama
  - University of California, Irvine Medical Center, Orange, California
  - Yale University School of Medicine, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was prematurely randomized while failing screening eligibility. This subject was counted in both 'Screen Failures' and 'Randomized Subjects/ITT population', leading to a discrepancy between the Enrollment number in the Protocol Section (27) and the number of participants Started in the Participant Flow module (26).
Groups:
- Treatment Group 1: Aprepitant Injectable Emulsion: Aprepitant injectable emulsion, 130 mg once daily (QD) for 14 days.
- Treatment Group 2: Placebo: Saline Placebo, QD for 14 days.
Period: Overall Study
Arm/Group | Treatment Group 1: Aprepitant Injectable Emulsion | Treatment Group 2: Placebo
Started | 12 | 14
Completed | 12 | 11
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Screen Failure | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population.
Groups:
- Treatment Group 1: Aprepitant Injectable Emulsion: Aprepitant injectable emulsion, 130 mg QD for 14 days.
- Total: Total of all reporting groups
Arm/Group | Treatment Group 1: Aprepitant Injectable Emulsion | Treatment Group 2: Placebo | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 10 | 16
  >=65 years | 6 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (15.64) | 57.7 (11.93) | 59.7 (13.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 13 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Alive and Discharged From the Hospital.
Description: ITT Population.
Time Frame: 14 Days.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1: Aprepitant Injectable Emulsion | Treatment Group 2: Placebo
Number analyzed (Participants) | 12 | 14
Participants | 11 | 10

2. Secondary Outcome: Time to Death or Respiratory Failure, Defined as Any of the Following: Endotracheal Intubation and Mechanical Ventilation; Oxygen Delivered by High-flow Nasal Cannula; Noninvasive Positive Pressure Ventilation; Extracorporeal Membrane Oxygenation (ECMO).
Time Frame: 56 Days.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment Group 1: Aprepitant Injectable Emulsion | Treatment Group 2: Placebo
Number analyzed (Participants) | 12 | 14
days | NA [2.00 to NA] — The number of subjects with death or respiratory failure was too small to estimate the median | NA [4.00 to NA] — The number of subjects with death or respiratory failure was too small to estimate the median

3. Secondary Outcome: Time to Discharge From Hospital.
Time Frame: 56 Days.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment Group 1: Aprepitant Injectable Emulsion | Treatment Group 2: Placebo
Number analyzed (Participants) | 12 | 14
days | 6.0 [3.00 to 8.00] | 8.0 [4.00 to 11.00]

4. Secondary Outcome: Change From Baseline in Interleukin 6 (IL-6).
Time Frame: Days 7, 14, 28, Discharge (from 2 to 43 days; median 6 days (Aprepitant), 8 days (Placebo))
Population: Overall Number of Participants Analyzed reflects the Total Enrolled ITT Population whereas Number Analyzed in each row reflects the number of subjects with IL-6 data reported at the specified timepoint.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Treatment Group 1: Aprepitant Injectable Emulsion | Treatment Group 2: Placebo
Number analyzed (Participants) | 12 | 14
pg/mL
  Baseline: number analyzed (Participants) | 11 | 12
  Baseline | 18.77 (26.321) | 19.11 (30.098)
  Day 7: number analyzed (Participants) | 4 | 8
  Day 7 | -27.98 (42.493) | 14.83 (65.384)
  Day 14: number analyzed (Participants) | 1 | 3
  Day 14 | 124.00 (NA) — The standard deviation is not defined when the sample size is equal to 1. | 204.30 (407.244)
  Day 28: number analyzed (Participants) | 1 | 1
  Day 28 | -8.00 (NA) — The standard deviation is not defined when the sample size is equal to 1. | 2.90 (NA) — The standard deviation is not defined when the sample size is equal to 1.
  Discharge: number analyzed (Participants) | 8 | 6
  Discharge | -17.41 (30.754) | -9.68 (18.107)

5. Secondary Outcome: Incidence of Treatment-emergent Adverse Events.
Description: Number of subjects reporting at least on Treatment-Emergent Adverse Event. Subjects reporting more than one event are counted only once using the highest severity.
Time Frame: Through Day 56
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1: Aprepitant Injectable Emulsion | Treatment Group 2: Placebo
Number analyzed (Participants) | 12 | 13
Participants | 8 | 5

ADVERSE EVENTS:
Time Frame: Through Day 56.
Description: One subject was prematurely randomized while failing screening eligibility. This subject was counted in both 'Screen Failures' and 'Randomized Subjects/ITT population'. ITT Population includes all subjects who are randomized. Safety Population includes all subjects who received at least one dose of any study drug (including placebo). All-Cause Mortality was assessed in the ITT population. Serious and Other Adverse Events were assessed in the Safety Population.
Arm/Group | Treatment Group 1: Aprepitant Injectable Emulsion | Treatment Group 2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 1/14
Serious Adverse Events (participants affected / at risk) | 2/12 | 2/13
Other Adverse Events (participants affected / at risk) | 8/12 | 5/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group 1: Aprepitant Injectable Emulsion (N=12) | Treatment Group 2: Placebo (N=13)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sinus node dysfunction (Cardiac disorders) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group 1: Aprepitant Injectable Emulsion (N=12) | Treatment Group 2: Placebo (N=13)
Candida infection (Infections and infestations) | 1 | 0
Leuconostoc infection (Infections and infestations) | 0 | 1
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 2
Tongue discomfort (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Candida test positive (Investigations) | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Study was terminated early by Heron, and was not terminated for safety reasons. The data reported is only safety data generated from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT04470622/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT04470622/SAP_001.pdf